CLINICAL TRIAL: NCT01892098
Title: Supplemental Zinc and Bone Turnover in Early Pubertal Females
Brief Title: Zinc and Bone Turnover Study in Adolescent Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R03HD054630 (NIH)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Bone; Growth; Osteoporosis
Keywords: Zinc; Bone; Adolescents; Growth
MeSH Terms: conditions — Osteoporosis | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc Sulfate (Active Comparator): Subjects enrolled in this arm will receive 9mg elemental zinc (23mg zn sulfate)/day for 4 weeks.
  Interventions: Dietary Supplement: Zinc Sulfate
- Cellulose Pill (Placebo Comparator): Subject enrolled in this arm will receive a placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc Sulfate — 9mg elemental zinc via 23mg zinc sulfate/day
  Arms: Zinc Sulfate
Dietary Supplement: Placebo — Cellulose pill given as placebo
  Arms: Cellulose Pill

SUMMARY:
The purpose of the study is to determine the effects of zinc supplementation on bone growth over four weeks. Participants will agree to attend two visits to our laboratory and at each will complete blood and urine samples, questionnaires related to diet and physical activity and will receive a bone scan at the first appointment.

DETAILED DESCRIPTION:
Significant accomplishments have been achieved with respect to our understanding of calcium and vitamin D and skeletal health, yet a body of scientific evidence has also identified understudied nutrients that have potential for reducing the burden of osteoporosis. Zinc has important roles in bone metabolism and there are indications from animal and human studies that beyond correcting skeletal and growth impairments under deficiency conditions, supplementation with zinc may have a bone health-promoting role. It has been postulated that the action of zinc on bone metabolism is partially mediated by Insulin-like growth factor one (IGF-I). Prior to undertaking a long-term bone trial, a short-term zinc supplementation trial is proposed to first determine if zinc alters intermediate markers of bone metabolism in healthy, early pubertal females (9-10.5 years of age). We hypothesize that healthy females receiving 24 mg zinc /day over 4 weeks will have elevated serum markers of bone formation and plasma growth factors compared to those receiving placebo. We further hypothesize that the differences between the zinc and placebo groups will vary by race. To test these hypotheses, we will screen early pubertal females to assure similar maturational status and conduct a 3-week, randomized, double-blind, placebo-controlled trial with a zinc supplementation (zinc sulfate; n=80) and a placebo (n=80) arm. The groups will be further divided by race (non-Hispanic White and non-Hispanic Black; n=40 per group). The specific aims are to determine if early pubertal females supplemented with zinc compared to those receiving placebo will have: 1) greater increases in markers of bone turnover favoring bone formation; 2) greater increases in plasma IGF-1 and IGFBP-3; and 3) changes in bone turnover markers, IGF-1 and IGFBP-3 that differ by race. In addition, anthropometric measures, maturity offset, sexual maturation, erythrocyte superoxide dismutase activity, ceruloplasmin, dietary intakes and physical activity will be determined. Findings from this study will provide preliminary evidence of whether supplementation with zinc is a viable nutrition strategy to improve biochemical indices of bone turnover and growth factors in young females. Moreover, the results will help determine if a long-term clinical bone trial is warranted to more definitely assess the potential for supplemental zinc to reduce the risk for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Female
* Ages 9-11
* Pre-menarchal
* Caucasian or African American

Exclusion Criteria:

* Menses
* Disease known to affect bone
* Drugs known to affect bone
* Vitamin/mineral supplements

Ages: 9 Years to 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2007-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Serum Zinc | 4 weeks
  Serum Zinc will be measured at the Baseline and 4 week time point to determine effects of placebo vs. supplement.
Plasma IGF-1 and IGFBP-3 | 4 weeks
  Plasma IGF-1 and IGFBP-3 will be measured at Baseline and 4-weeks and analyzed using ELISA to determine changes.
procollagen type 1 amino-terminal propeptide (P1NP) | 4 weeks
  Bone turnover marker procollagen type 1 amino-terminal propeptide,

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Lewis, PhD, Principal Investigator — The University of Georgia

REFERENCES:
- [Derived] Lobene AJ, Kindler JM, Jenkins NT, Pollock NK, Laing EM, Grider A, Lewis RD. Zinc Supplementation Does Not Alter Indicators of Insulin Secretion and Sensitivity in Black and White Female Adolescents. J Nutr. 2017 Jul;147(7):1296-1300. doi: 10.3945/jn.117.248013. Epub 2017 Jun 7. PMID 28592518
- [Derived] Kindler JM, Pollock NK, Laing EM, Jenkins NT, Oshri A, Isales C, Hamrick M, Lewis RD. Insulin Resistance Negatively Influences the Muscle-Dependent IGF-1-Bone Mass Relationship in Premenarcheal Girls. J Clin Endocrinol Metab. 2016 Jan;101(1):199-205. doi: 10.1210/jc.2015-3451. Epub 2015 Nov 17. PMID 26574958
- [Derived] Berger PK, Pollock NK, Laing EM, Chertin V, Bernard PJ, Grider A, Shapses SA, Ding KH, Isales CM, Lewis RD. Zinc Supplementation Increases Procollagen Type 1 Amino-Terminal Propeptide in Premenarcheal Girls: A Randomized Controlled Trial. J Nutr. 2015 Dec;145(12):2699-704. doi: 10.3945/jn.115.218792. Epub 2015 Oct 21. PMID 26491117